CLINICAL TRIAL: NCT02078193
Title: An Exploratory, Open-label, Single Center Study to Assess the Efficacy of NULOJIX (Belatacept) in Reducing Donor Specific Human Leukocyte Antigen (HLA) Antibody (DSA) Strength in Maintenance Kidney Transplant Recipients
Brief Title: Efficacy of Belatacept in Reducing DSA
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: East Carolina University (Other)
Responsible Party: Principal Investigator, Paul Bolin, Dr. Paul Bolin, MD, East Carolina University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IM103-302
Record Dates: First submitted 2014-03-03; First posted 2014-03-05 (Estimated); Results first posted 2017-07-06 (Actual); Last update posted 2017-08-01 (Actual); Status verified 2017-07

CONDITIONS: Kidney Transplantation
MeSH Terms: interventions — Abatacept

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Belatacept (Experimental): Participants will be converted from their current MMF to once a month infusions of Belatacept
  Interventions: Drug: Belatacept

INTERVENTIONS:
Drug: Belatacept — Patients will be converted from their MMF to Belatacept

SUMMARY:
The primary objective of this study is to demonstrate that administration of belatacept in maintenance kidney transplant recipients may cause a reduction in Donor Specific HLA Antibody (DSA).

DETAILED DESCRIPTION:
The aim of this study is to evaluate patients converted to belatacept in combination with Mycophenolate Mofetil (MMF) with corticosteroids with respect to their DSA titer. Patients in this study will be converted from their calcineurin inhibitor (CNI) to belatacept from baseline in an attempt to down-modulate antibody production by B-cells. Dosing will be calculated per prescribing information for dosing maintenance phase (5mg per kg every 28 days.

ELIGIBILITY:
Inclusion Criteria:

* Recipients of cadaveric, living related or living unrelated kidney transplant with positive DSA titer (two positive tests) and enrolled within 6 months of DSA detection.
* Patients with stable renal function. Stable renal function is defined as one serum creatinine (SCr) value that is +/- 10% of the baseline SCr within 3 months of enrollment (eGFR >/= 35 and </= 75 mL/min/1.73m^2).
* Patients who are EBV seropositive
* Males and females, 18-75 years of age;
* Patients currently receiving mycophenolic acid (MPA) (CellCept daily or myfortic daily), cyclosporine or tacrolimus with corticosteroids as part of their immunosuppressive regimen
* Patients willing to be converted to belatacept from cyclosporine or tacrolimus.
* Females of childbearing potential must have a negative pregnancy test prior to enrollment. The test should be performed at baseline visit. Effective contraception must be used during the trial, and for 4 weeks following discontinuation of the study medication;
* Patients who are willing and able to participate in the full course of the study and from whom written informed consent has been obtained.

Exclusion Criteria:

* Multi-solid or cellular organ transplants (e.g. combined with pancreas, liver, islet, bone marrow), either concurrent or previous (with exception that a second kidney transplant is allowed);
* Evidence of graft rejection or treatment of acute rejection within 14 days prior to Baseline visit;
* Patients who have received any investigational drug within 4 weeks prior to study entry;
* Patients with HLA identical
* Patients who are Epstein-Barr virus (EBV) seronegative
* Presence of clinically significant infection requiring continued therapy, chronic infection (e.g. HIV, Hep B and Hep C), malignancy (within last 5 years, except excised squamous or basal cell carcinoma of the skin), lymphoma or renal toxicity that would interfere with the appropriate conduct of the study;
* Evidence of severe liver disease (incl. abnormal liver profile i.e. Aspartate Aminotransferase (AST), Alanine Aminotransferase (ALT) or total bilirubin >/= 3 times ULN) or severe diarrhea or active peptic ulcer disease that would interfere with the appropriate conduct of the study;
* Abnormal physical or laboratory findings of clinical significance within 2 weeks of inclusion which would interfere with the objectives of the study;
* Patients with symptoms of significant somatic or mental illness or evidence of drug and/or alcohol abuse;
* Patients receiving > 10 mg/day prednisone dose;
* History of hypersensitivity to any of the study drugs or to drugs with similar chemical structures to belatacept;
* Patients not making DSA antibodies;
* Pregnant or nursing (lactating) women, where pregnancy is defined as the state of a female after conception and until the termination of gestation, confirmed by a positive human chorionic gonadotropin (hCG) laboratory test (local); females of childbearing potential who are unwilling to use effective study-approved contraceptives and who are planning to become pregnant; Sexually active fertile men must use effective birth control if their partners are women of child bearing potential;
* Any other medical condition that, in the opinion of the site investigator based on recall or chart review would interfere with completing the study, including but not limited to visual problems or cognitive impairment.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2013-11; Primary Completion 2016-07 (Actual); Study Completion 2016-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Paul Bolin, MD, Principal Investigator — East Carolina University, Department Chair of Internal Medicine
Locations (1):
- East Carolina University, Greenville, North Carolina, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Belatacept: All patients enrolled will be converted to Belatacept from prograf.
Period: Overall Study
Arm/Group | Belatacept
Started | 3
Completed | 3
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Belatacept
Number analyzed (Participants) | 3
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.3 (5.51)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 2
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 3

OUTCOME MEASURES:

1. Primary Outcome: Change of Donor Specific Antibodies (DSA)
Description: DSA levels will be measured using microbeads coated with Class I or Class II human leukocyte antigens (HLA) and read using a Luminex flow cytometer. Participants will be converted from their current Mycophenolate Mofetil (MMF) to once a month infusions of Belatacept.
Time Frame: one year
Measure: Mean (Standard Deviation); unit: percent change in DSAs
Groups:
- Belatacept: Participants will be converted from their current Mycophenolate Mofetil (MMF) to once a month infusions of Belatacept
  Belatacept: Patients will be converted from their MMF to Belatacept
Arm/Group | Belatacept
Number analyzed (Participants) | 3
percent change in DSAs | 35.7 (45.8)

2. Secondary Outcome: Safety
Description: Incidence of infections
Time Frame: one year
Population: Number of participants with infections
Measure: Number; unit: Participant
Groups:
- Belatacept: Participants who received Belatacept by IV infusion.
Arm/Group | Belatacept
Number analyzed (Participants) | 3
Participant | 2

3. Other Pre Specified Outcome: Number of Participants With Chronic Kidney Rejection
Description: Incidence of chronic kidney rejection
Time Frame: One year
Measure: Number; unit: participants
Arm/Group | Belatacept
Number analyzed (Participants) | 3
participants | 0

ADVERSE EVENTS:
Arm/Group | Belatacept
All-Cause Mortality (participants affected / at risk) | 0/3
Serious Adverse Events (participants affected / at risk) | 0/3
Other Adverse Events (participants affected / at risk) | 2/3
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Belatacept (N=3)
COPD exacerbation (Respiratory, thoracic and mediastinal disorders) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No